CLINICAL TRIAL: NCT00767936
Title: Viral and Host Factors Associated With Development of Hepatitis B Virus-related Hepatocellular Carcinoma
Brief Title: Viral & Host Factors Associated With Hepatitis B Virus-related Hepatocellular Carcinoma
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: HEP0013; 98795 (Other: Stanford University Alternate IRB Approval Number); SU-05222008-1183 (Other: Stanford University); NCT00767936
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Liver Cancer; Hepatitis B; Hepatitis C; Hepatobiliary Cancers Liver; Hepatobiliary Cancers
MeSH Terms: conditions — Liver Neoplasms; Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood

SUMMARY:
Adult liver cancer is the third leading cause of cancer deaths worldwide. The major risk factor for liver cancer is hepatitis B virus (HBV) infection. The purpose of the study is to sequence the HBV genome in patients with chronic HBV infection, and in patients with liver cancer resulting from chronic HBV infection. The goal is to identify mutations in the HBV genome that predisposes these high risk individuals to the development of liver cancer.

ELIGIBILITY:
Inclusion Criteria:1. Patients diagnosed with liver cancer based on biopsy or serum AFP level, associated with characteristic hypervascular liver tumors on triphasic spiral CT scan or MRI.

2. Patients with non-cancer liver conditions such as cirrhosis, adenoma, cholangioma, or nodular hyperplasia.

3. Patients with hepatitis B or hepatitis C viral infections not associated with liver cancer. Exclusion Criteria:No other patients except those listed above will be recruited. Additionally, patients will be excluded if, upon looking through their medical records, information required for data analysis are missing.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver cancer and non-cancer liver conditions
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2008-03; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
identify mutations in the hepatitis B virus genome that predisposes these high risk individuals to the development of liver cancer | one time
  We will be using blood specimens collected through another protocol

CONTACTS AND LOCATIONS:
Overall Officials: Samuel So, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States